CLINICAL TRIAL: NCT03369587
Title: Handwriting Interventions for People With Parkinson's
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not feasible to restarted after Covid pandemic - analysis will be on data collected before study suspended
Sponsor: Oxford Brookes University (Other)
Collaborators: European Parkinson's Therapy Centre (Unknown)
Responsible Party: Principal Investigator, Dr Johnny Collett, Senior Research Fellow, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 171073
Record Dates: First submitted 2017-07-18; First posted 2017-12-12 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: Handwriting, Micrographia
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A phase II exploratory randomised controlled trial of a handwriting intervention with an active comparator control group and blinded assessments
Who Masked: Outcomes Assessor
Masking Description: Assessor Blind to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diverging lines (Experimental): What: Handwriting practice at home delivered through handwriting workbooks. The workbook consists of diverging lines. Participants will be instructed to write a daily diary (a reflection of their day) aiming for letters letter size to be consistent with the lines. Participant will be instructed to take a long as they need to complete the daily diary and focus and concentrate the handwriting and achieving the size dictated by the lines. They will be asked to do this daily, but at least 5 days a week for 6 weeks. Tailoring and progression: The nature of the handwriting program is that it accounts for individual ability; participant will be asked to write as much as they can during the practice session, whilst concentrating on their handwriting.
  Interventions: Behavioral: Handwriting Practice
- Parallel lines (Active Comparator): What: Handwriting practice at home delivered through handwriting workbooks. The workbook consists of parallel lines. Participants will be instructed to write a daily diary (a reflection of their day) aiming for letters letter size to be consistent with the lines. Participant will be instructed to take a long as they need to complete the daily diary and focus and concentrate the handwriting and achieving the size dictated by the lines. They will be asked to do this daily, but at least 5 days a week for 6 weeks. Tailoring and progression: The nature of the handwriting program is that it accounts for individual ability; participant will be asked to write as much as they can during the practice session, whilst concentrating on their handwriting.
  Interventions: Behavioral: Handwriting Practice

INTERVENTIONS:
Behavioral: Handwriting Practice — Self-directed home handwriting practice daily for 6 weeks

SUMMARY:
Background: Problems with handwriting are frustrating and debilitating and affect the majority of people with Parkinson's. Manifest as micrographia it is a distinctive feature of the condition characterised by small handwriting and/or a progressive reduction in size through a sentence[2] coupled with a reduction in writing speed and legibility.

In Parkinson's impaired automaticity is thought to contribute to handwriting deficits and attention has been shown to improve both 'consistent' (small handwriting) and 'progressive' (progressive reduction in letter size through a sentence) aspects of the symptom. Moreover, recent interventional studies indicate handwriting may be improved through practice. This study is investigating a novel handwriting practice stimulus to improve symptoms of micrograpthia

Question: Is a diverging line cued handwriting intervention potentially more effective at improving symptoms of mircograpthia than a parallel line cued handwriting intervention in people with Parkinson's?

Specifically, an assessor blind randomised controlled exploratory trial will:

1. Estatimate the effect of the intervention on measures of: Handwriting amplitude (consistent and progressive reduction), hand writing performance and percieved handwriting difficulties.
2. Explore the appropriateness of these outcome measures
3. Explore the approriateness of eligibilty criteria
4. Explore intervention fidelity
5. Explore participants views of the intervention

Design: A phase II exploratory randomised controlled trial of a handwriting intervention with an active comparator control group and blinded assessments

Setting: The intervention will be carried out at home

Sample size: This study is not designed to determine efficacy. The aim to recruit a total of 50 people (25 people per group) in order to estimate the effects on outcome measures and achieve the aims of this exploratory trial.

Assessment: Participants will be asked to follow their usual Parkinson's medication regime and if they have ON and OFF periods, assessments will be carried out during ON state.

Duration and follow-up: the assessment is schedule 0Weeks (baseline), 6weeks (end intervention) and 12weeks (follow up). Assessments will be carried out by a researcher blind to trial arm allocation using all outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Diagnosis of idiopathic Parkinson's disease
* A score of ≤3 on the Hoehn and Yahr scale
* Self-reported problem with handwriting (≥1 UPDRSII, 2.7)
* Able to communicate in Italian
* Following a stable medication regimen (no changes in the last 2 weeks and anticipated changes for the course of the study).

Exclusion Criteria:

* Severe depression or psychosis (history of),
* reduced cognition that would preclude active involvement or capacity to consent (according to stages outlined in metal capacity act (ie trigger, information, existing diagnosis, functional test))
* Orthopaedic, neurological or other condition that significantly impairs hand function,
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Micrograpthia: Area of 'el' 8 character text sequence writing task | 6 weeks
  Area (maximum height x maximum width) of handwritten cursive 'elelelel' character sequence measured to the nearest of 0.5mm
Self-reported problem with handwriting: Item 2.7 on the Movement Disorders Society Unified Parkinson's Rating Scale | 6 weeks
  A scale from 0-4 (0: normal: no problems, 4: severe: most or all words cannot be read) asking 'Over the past week, have people usually had trouble reading your handwriting?'
Writing speed: Time taken to write an Italian proverb | 6 weeks
  Time taken to the nearest 10th second to hand write the sentence (written across one line): 'Chi lascia la via vecchia per la nuova, sa quello che lascia ma non sa quello che trova'
Writing amplitude: Area of the both 'lascia' contained in an Italian proverb | 6 weeks
  Area (maximum height x maximum width) of 'lascia' contained in handwritten sentence: 'Chi lascia la via vecchia per la nuova, sa quello che lascia ma non sa quello che trova'. Measured to the nearest 0.5mm

SECONDARY OUTCOMES:
Micrograpthia under cognative motor interference: Area of 'el' 8 character text sequence writing task | 6 weeks
  Area (maximum height x maximum width) of handwritten cursive 'elelelel' character sequence performed concurrently with cognative task (serial 3 subtraction). Measured to the nearest of 0.5mm
Micrograpthia under cognative motor interference: Area of 'el' 8 character text sequence writing task | 12 weeks
  Area (maximum height x maximum width) of handwritten cursive 'elelelel' character sequence performed concurrently with cognative task (serial 3 subtraction). Measured to the nearest of 0.5mm
Legibility of Free writing | 6 weeks
  Ratio between total number of words written and total number of legible words written during a 5 minutes of free writing task: A reflection on the day
Legibility of Free writing | 12 weeks
  Ratio between total number of words written and total number of legible words written during a 5 minutes of free writing task: A reflection on the day
EQ-5D-5L | 6 weeks
  Standardized Instrument to measure health outcome
EQ-5D-5L | 12 weeks
  Standardized Instrument to measure health outcome
Micrograpthia: Area of 'el' 8 character text sequence writing task | 12 weeks
  Area (maximum height x maximum width) of handwritten cursive 'elelelel' character
Self-reported problem with handwriting: Item 2.7 on the Movement Disorders Society | 12 weeks
  0-4 scale (0: normal: no problems, 4: severe: most or all words cannot be read) asking 'Over the past week, have people usually had trouble reading your handwriting?'
Writing speed: Time taken to write an Italian proverb | 12 weeks
  Time taken to the nearest 10th second to hand write the sentence (written across one line): 'Chi lascia la via vecchia per la nuova, sa quello che lascia ma non sa quello che trova'
Writing amplitude: Area of the both 'lascia' contained in an Italian proverb | 12 weeks
  Area (maximum height x maximum width) of 'lascia' contained in handwritten sentence: 'Chi lascia la via vecchia per la nuova, sa quello che lascia ma non sa quello che trova'. Measured to the nearest 0.5mm

CONTACTS AND LOCATIONS:
Locations (1):
- European Parkinson's therapy centre, Darfo Boario Terme, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided